CLINICAL TRIAL: NCT05226468
Title: A 2-part, First-in-patient, Open-label, Dose-escalation and Expansion Cohort Study of NEI-01 as Monotherapy in Patients With Advanced Solid Tumors or Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: An Early Phase Study of NEI-01 in Patients With Solid Tumors or Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New Epsilon Innovation Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEI01-20001
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: 3+3 design for dose escalation in Part 1 and Simon's optimal two stage design for dose expansion in Part 2.
  NEI-01 as single agent in both Part 1 and Part 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEI-01 (Experimental): Single Arm
  Interventions: Drug: NEI-01

INTERVENTIONS:
Drug: NEI-01 — Part1:
  Single dose period: Intravenous single dose of NEI-01 with 4 ascending dose levels.
  Multiple dose period: Intravenous weekly dose of NEI-01 for 9 weeks with 4 ascending dose levels.
  Part2:
  Intravenous weekly dose of NEI-01 at the recommended dose obtained from Part 1

SUMMARY:
This is an early phase clinical study using NEI-01 as single agent in oncology indication. This is an open label study and it's divided into two parts.

Part 1: This part is ascending dose design to determine the safety and tolerability of NEI-01 and find out recommended dose of NEI-01 in solid tumor patient.

Part 2: This part is extended dose design to determine the effectiveness of NEI-01 in in solid tumor and acute myeloid leukemia patients.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, 2-part dose-escalation and cohort expansion study of NEI-01 monotherapy in patients with advanced solid tumors or relapsed/refractory acute myeloid leukemia (AML).

This study consists of 2 parts: Part 1) the dose-escalation part in patients with advanced solid tumors and Part 2) the cohort expansion part of the study of NEI-01 in patients with advanced solid tumors or relapsed/refractory AML.

The primary objective of Part 1 are to evaluate the safety and tolerability of NEI-01, identify the maximum tolerated dose (MTD), and define the RDL for Part 2 of the study. The pharmacokinetics (PK) profile and preliminary efficacy of NEI-01 will also be evaluated whereas Part 2 is to assess the safety, tolerability and efficacy at weekly doses of NEI-01 at the RDL in subjects with advanced solid tumors or relapsed/refractory AML.

Part 1: This part will be conducted in 4 dose ascending cohorts, including single dose and multiple dose periods. The DLT will be observed up to pre-dose assessment of Day 50. Dose escalation decision will be made based on safety data collected from all the subjects enrolled in the dose group will be evaluated by a Data and Safety Monitoring Committee (DSMC).

Part 2: This part will only include the recommended dose (RDL) defined in Part 1. NEI-01 will be administered as a single agent in patients with advanced solid tumors (Cohort 1) or relapsed/refractory AML (Cohort 2). It will start after the RDL has been defined in Part 1 of the study. All subjects will receive weekly doses of NEI-01 at the RDL.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be capable of giving written informed consent.
2. Confirmed diagnosis of advanced solid tumor or relapsed/refractory AML as detailed below:

   1. For Part 1 and 2 (Cohort 1): Histologically or cytologically confirmed diagnosis of any locally advanced or metastatic solid tumor
   2. For Part 2 (Cohort 2): Histologically or cytologically confirmed diagnosis of relapsed or refractory AML as defined by World Health Organisation (WHO) classification
3. Existence of all of the following medical conditions or diagnoses:

   For Solid Tumor Population:
   1. At least one measurable target lesion at screening, as defined by RECIST 1.1;
   2. Life expectancy ≥ 12 weeks at screening;
   3. ECOG performance status of 0 or 1 at screening;
   4. Adequate bone marrow function at screening, as defined by: Hb ≥ 8 g/dL; ANC ≥ 1.5 × 109/L; AND Platelet count ≥ 75× 109/L;
   5. Adequate coagulation function at screening, as defined by: PT or INR ≤ 1.5 × ULN; AND aPTT ≤ 1.5 × ULN;
   6. Adequate liver function at screening, as defined by: Total bilirubin ≤ 1.5 × ULN; AND AST and ALT ≤ 2.5 × ULN OR ≤ 5 × ULN;
   7. Adequate renal function at screening, as defined by: Creatinine ≤ 1.5 × ULN; OR Creatinine clearance ≥ 50 mL/min.

   For Part 2 (Cohort 2) - AML Population:
   1. Life expectancy ≥ 12 weeks at screening;
   2. ECOG performance status ≤ 2 at screening;
   3. Adequate liver function at screening, as defined by: Total bilirubin ≤ 1.5× ULN; AND AST and ALT ≤ 3 ULN;
   4. Adequate renal function at screening, as defined by: Creatinine ≤ 1.5 × ULN; OR Creatinine clearance ≥ 30 mL/min (by the Cockcroft Gault method).
4. Willingness and agreement to undertake measures to avoid pregnancy of the subject or the subject's sexual partner(s)
5. A female subject must be willing and agree to avoid engagement in breastfeeding.
6. Willingness and agreement to avoid blood donation.

Exclusion Criteria:

1. History of any of the following diseases or conditions:

   1. Previous or concurrent active cancer that is distinct in primary site or histology from the cancer being evaluated in this study;
   2. Known CNS metastasis(es), unless the metastasis(es) was/were treated and became stable and the subject does not require systemic corticosteroids for management of CNS symptoms for at least 14 days prior to the first dose of study intervention;
   3. Any history of or current active cardiac disease or dysfunction;
   4. Known history of HIV infection;
   5. Known history of active HBV infection;
   6. Known history of active HCV infection.
2. Existence of any of the following medical conditions or diagnoses:

   1. Positive pregnancy test;
   2. Active infection requiring treatment by systemic therapy;
   3. Any unresolved toxicity related to any prior therapy of ≥ Grade 2 (as defined by NCI CTCAE v5.0) prior to the first dose of the study intervention.
3. Use of any of the following prior or concomitant medications, therapies or interventions:

   1. Prior treatment with ADI-PEG-20 or another experimental arginine deprivation strategy;
   2. Any anti-cancer therapy within 21 days prior to the first dose of the study intervention and/or during the subject's participation in the study;
   3. Any surgery within 28 days prior to the first dose of the study intervention.
4. Prior or concurrent participation in any other clinical study
5. Any clinically significant concomitant disease or condition that, in the reasonable opinion of the investigator, may interfere with the subject's participation in this study or pose an unacceptable safety risk for the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Part1: MTD / RDL | 12 months
  MTD (Maximum tolerable dose) / Recommended dose level (RDL)
Part1: Occurrence of DLT | Day 1 of single dosing till pre-dose assessment of Day 50
  Occurrence of DLT (Dose Limiting Toxicity)
Part1: Occurrence of AE and SAE（NCI CTCAE 5.0） | From start of study until 28 days after last dose
  Occurrence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part1: Frequency of AE and SAE（NCI CTCAE 5.0） | Time Frame: From start of study until 28 days after last dose
  Frequency of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part2: Occurrence of AE and SAE（NCI CTCAE 5.0） | From start of study until 28 days after last dose
  Occurrence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part2: Frequency of AE and SAE（NCI CTCAE 5.0） | From start of study until 28 days after last dose
  Frequency of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part 2: DCR | From prior to first dose of study medication, within 2 days after Week 6 Day 1, then every 6 weeks until treatment discontinuation
  Disease Control Rate (DCR) Evaluate by RECIST 1.1 or 2003 IWG AML Response Criteria

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics Profile - AUC 0-t | Single dose : Pre-dose, 0 hour, 0.25hour, 0.5hour, 0.75 hour, 1hour, 6hours, 12hours, 24hours, 48hours, 72 hours, 168 hours, 336 hours and 504 hours post-end of infusion of the initial dose
  The area under the plasma drug concentration-time curve up to t = 504h (AUC0-t)
Part 1: Pharmacokinetics Profile - AUC 0-infinity | Single dose : Pre-dose, 0 hour, 0.25hour, 0.5hour, 0.75 hour, 1hour, 6hours, 12hours, 24hours, 48hours, 72 hours, 168 hours, 336 hours and 504 hours post-end of infusion of the initial dose
  The area under the plasma drug concentration-time curve to infinite time (AUC0-infinity)
Part 1: Pharmacokinetics Profile - Cmax | Single dose : Pre-dose, 0 hour, 0.25hour, 0.5hour, 0.75 hour, 1hour, 6hours, 12hours, 24hours, 48hours, 72 hours, 168 hours, 336 hours and 504 hours post-end of infusion of the initial dose
  The maximum plasma concentration (Cmax)
Part 1: Pharmacokinetics Profile - Ctrough | Multiple dose: Pre-dose, 0.25hour post-end of infusion of Week 1 Day 1 (W1D1), W2D1, W3D1, W4D1 and W5D1
  The trough level of observed plasma concentration (Ctrough)
Part 1: Pharmacokinetics Profile - Cpeak | Multiple dose: Pre-dose, 0.25hour post-end of infusion of Week 1 Day 1 (W1D1), W2D1, W3D1, W4D1 and W5D1
  The peak level of observed plasma concentration (Cpeak)
Part 1: DCR | From prior to first dose of study medication, within 2 days after Week 6 Day 1, then every 6 weeks until treatment discontinuation, an average of 9 months
  Disease Control Rate (DCR) Evaluate by RECIST 1.1
Part 2: ORR | From prior to first dose of study medication, within 2 days after Week 6 Day 1, then every 6 weeks until treatment discontinuation, an average of 9 months
  Objective Response Rate (ORR) Evaluate by RECIST 1.1 or 2003 IWG AML Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kwok, PhD, Study Director — New Epsilon Innovation Limited
Locations (1):
- The University of Hong Kong Phase I Clinical Trials Centre, Hong Kong, Hong Kong